CLINICAL TRIAL: NCT04120883
Title: Oral Hydroxychloroquine for Retinitis Pigmentosa Caused by P23H-RHO (Substitution of Proline to Histidine at Codon 23 of the Rhodopsin Protein)
Brief Title: Oral Hydroxychloroquine (HCQ) for Retinitis Pigmentosa Caused by P23H- Rhodopsin (RHO)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to recruit additional participants after multiple extensions to planned enrollment period.
Sponsor: University of Michigan (Other)
Collaborators: Cures Within Reach (Other)
Responsible Party: Principal Investigator, David Zacks, Professor of Ophthalmology and Visual Sciences, University of Michigan
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00164470
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Retinitis Pigmentosa
Keywords: P23H-RHO; eye disease
MeSH Terms: conditions — Retinitis Pigmentosa; Eye Diseases | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: The start of intervention for treatment arm 2 of the study will be delayed until preliminary safety of the drug is established with the 6 patients in treatment arm 1 at the first follow-up visit (4 months).
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HCQ treatment 1 (Experimental): In treatment arm 1, the dose of study drug will be 4 mg/kg/day. The daily dose will not exceed 400 mg. In both groups, the dose will be rounded down to 100, 200, 300, or 400 mg/day.
  Interventions: Drug: Hydroxychloroquine lower dose
- HCQ treatment 2 (Experimental): In treatment arm 2, the dose of the study drug will be 5 mg/kg/day. The daily dose will not exceed 400 mg. In both groups, the dose will be rounded down to 100, 200, 300, or 400 mg/day.
  Interventions: Drug: Hydroxychloroquine higher dose

INTERVENTIONS:
Drug: Hydroxychloroquine lower dose — The participants weight will be measured and converted to kilograms. The participants will receive 4 mg/kg/day. At the first follow-up visit (4 months) weight will be re-measured and the study drug dosing will be adjusted accordingly if the dosing has changed. Participants receiving 100 mg daily will be instructed to ingest one 200 mg tablet every other day. Participants receiving 200 mg daily will be instructed to ingest one 200 mg tablet daily. Participants receiving 300 mg daily will be instructed to alternate days ingesting two 200 mg tablets and one 200 mg tablet. Participants receiving 400 mg daily will be instructed to ingest two 200 mg tablets daily.
  Other Names: plaquenil
  Arms: HCQ treatment 1
Drug: Hydroxychloroquine higher dose — The start of intervention for treatment arm 2 of the study will be delayed until preliminary safety of the drug is established with the 6 patients in treatment arm 1 at the first follow-up visit (4 months).
  The participants in this group will receive 5 mg/kg/day. At the first follow-up visit (4 months) weight will be re-measured and the study drug dosing will be adjusted accordingly if the dosing has changed. Participants receiving 100 mg daily will be instructed to ingest one 200 mg tablet every other day. Participants receiving 200 mg daily will be instructed to ingest one 200 mg tablet daily. Participants receiving 300 mg daily will be instructed to alternate days ingesting two 200 mg tablets and one 200 mg tablet. Participants receiving 400 mg daily will be instructed to ingest two 200 mg tablets daily.
  Other Names: plaquenil
  Arms: HCQ treatment 2

SUMMARY:
This research study is being done to learn what effect 12 months of treatment with oral hydroxychloroquine (HCQ) will have on the retina in people with retinitis pigmentosa (RP). The hypothesis is that treatment with HCQ is safe and tolerable in patients with autosomal dominant retinitis pigmentosa (adRP) caused by P23H-RHO, and may arrest progression of retinal degeneration by altering the autophagy pathway in photoreceptors.

Participants that meet eligibility and agree to the study will be asked to take the study medication (HCQ) for 12 months and have evaluations for up to approximately 18 months from the baseline visit. There will be a total of 6 visits (1 is a phone visit) and will include general examinations, blood work, electrocardiograms, along with special testing of the retina.

ELIGIBILITY:
Inclusion Criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Signed and dated informed consent form
* Early Treatment Diabetic Retinopathy Study Best Corrected Visual Acuity (ETDRS BCVA) of 20 letters (approximately 20/400 Snellen) or better in at least one eye
* Clinical diagnosis of autosomal dominant retinitis pigmentosa
* Confirmed to have one copy of the P23H-RHO pathogenic variant by genetic testing at a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory
* Clarity of ocular media and adequate pupillary dilation to allow for adequate clinical ocular examination and retinal imaging
* Ability to perform testing required by the study as determined by the investigator
* Ability to take oral medication (medication tablets must be swallowed whole) and be willing to adhere to the daily medication regimen
* For females of reproductive potential: use of highly effective contraception beginning no later than 1 week after the first screening visit, and agreement to use such a method during study participation and through the end of the washout period (6 months after the end of HCQ administration)
* Agreement to adhere to Lifestyle Considerations throughout study duration (take the study drug with meals, avoid taking over-the-counter antacids or kaolin-containing products 4 hours before or after taking the study drug)

Exclusion Criteria:

* Use of any other drugs which are known to prolong the QT interval
* Concurrent use of any of the following drugs, if the drug cannot be discontinued or substituted: digoxin, antiepileptic medications, cimetidine, methotrexate, cyclosporine, praziquantel, ampicillin
* Current or previous use of tamoxifen
* Pregnancy or lactation
* Known allergy or hypersensitivity to hydroxychloroquine or any other 4-aminoquinoline drugs (chloroquine, amodiaquine, mefloquine, quinacrine, etc.), or known history of glucose-6-phosphate dehydrogenase deficiency
* Treatment with another investigational medical intervention for retinitis pigmentosa within 3 months, or any ever previous treatment with an investigational surgical intervention
* Any pre-existing cardiac, renal, hepatic, or hematologic disease, any prior history of psoriasis or porphyria, or any alcoholism
* Abnormal screening laboratory values including aspartate transaminase (AST) or alanine transaminase (ALT) > 2.0 x upper limit of normal, subnormal glomerular filtration rate (< 90 mL/min/1.73m2) or abnormal complete blood count attributable to underlying hematologic disease such as malignancy, aplastic anemia, agranulocytosis, leukopenia, or thrombocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Change in Ellipsoid zone area measured by Spectral-Domain Optical Coherence Tomography (SD-OCT) | screening up to 18 months
  These will be performed at: screening, baseline, 4 months, 12 months, and 18 months
Change in Retinal sensitivity (decibels) measured by scotopic and mesopic microperimetry | screening up to 18 months
  These will be performed at: screening, baseline, 4 months, 12 months, and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: David Zacks, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, individual participant data that underlie reported results will be shared.
Supporting Information: Study Protocol
Time Frame: Data be available beginning 9 months after publication and ending 36 months after publication.
Access Criteria: Researchers who provide a methodologically sound proposal can access the data. Types of analyses: to achieve proposed aims. Proposals should be directed to the study Principal Investigator. To gain access, data requestors will need to sign a data access agreement.